CLINICAL TRIAL: NCT06245954
Title: Learning Curve for the Diagnosis of Interstitial Lung Disease by Transbronchial Lung Cryobiopsy and the Role of Standardized Training in It
Brief Title: The Role of Standardized Training in the Diagnosis of Interstitial Lung Disease by Transbronchial Lung Cryobiopsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Gang Hou, Principal Investigator, China-Japan Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ZRJY2021-BJ08-03-02
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Transbronchial Lung Cryobiopsy
Keywords: transbronchial lung cryobiopsy; standardized training; learning curve; bronchoscopist

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standardized training group (Experimental): The bronchoscopists in this group will accept simulation training by means of simulators and extracorporeal lungs
  Interventions: Other: simulated training
- Traditional teaching model group (Other): The bronchoscopists in this group will accept traditional lectures, hands-on demonstrations and so on to learn TBLC
  Interventions: Other: traditional bedside teaching

INTERVENTIONS:
Other: simulated training — Simulation training of bronchoscopists by means of simulators and extracorporeal lungs
  Arms: Standardized training group
Other: traditional bedside teaching — TBLC training for bronchoscopists through traditional lectures, hands-on demonstrations
  Arms: Traditional teaching model group

SUMMARY:
The aim of this study was to conduct a prospective randomized controlled trial to design simulator and in vitro lung standardized training, to perform a learning curve evaluation of transbronchial lung cryobiopsy (TBLC) operating physicians, and to assess the role of standardized training in TBLC.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* suspected ILD.
* ≤3 months since HRCT
* Forced vital capacity (FVC) ≥50% of predicted value
* Diffused lung carbon monoxide (DLCO) ≥35% predicted value
* Echocardiography ≤ 12 months
* Estimated pulmonary artery systolic pressure ≤40 mmHg
* Body mass index (BMI) ≤35 kg/m2
* Patient consent for experimentation

Exclusion Criteria:

* Patients with platelet counts less than 50 × 109/L or prothrombin time international normalized ratio (INR) higher than 1.5
* Patients refused to participate in the experiment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Obtain pathologic quality assessment of specimens | 1 month
  The quality of TBLC sampling specimens was scored by two professional pathologists on a specialized pathology scale.
histopathological pattern diagnosis rate | 1 month
  Diagnosis of histopathological patterns was performed by two specialized pathologists to determine a consistent diagnostic rate.
diagnostic rate of multidisciplinary discussions | 1 month
  Diagnostic rates based on composite TBLC, BAL, clinical and imaging data in a multidisciplinary discussion by clinical experts

SECONDARY OUTCOMES:
Occurrence of short-term adverse events | 24 hours or 7 days
  bleeding and pneumothorax occurred with 24 hours after TBLC, acute exacerbation of ILD and death occurred with 7 days after TBLC

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China